CLINICAL TRIAL: NCT03919890
Title: A First-in-human, Randomised, Placebo-controlled, Double-blind, Single and Multiple Dose Study to Explore the Safety, Tolerability, PK and PD of Oral Doses of ONO-7684 in Healthy Subjects Under Fed and Fasted Conditions
Brief Title: A Two-Part Study to Assess the Safety, Tolerability, PK and PD of ONO-7684 in Healthy Adult Volunteers
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ono Pharmaceutical Co. Ltd (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Double | Purpose: Treatment
Other Study IDs: ONO-7684-01
Record Dates: First submitted 2019-03-14; First posted 2019-04-18 (Actual); Last update posted 2019-12-09 (Actual); Status verified 2019-12

CONDITIONS: Venous Thromboembolism
MeSH Terms: conditions — Venous Thromboembolism

STUDY DESIGN:
Who Masked: Participant, Investigator
Masking Description: Double-blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (6):
- ONO-7684 Part A1 (Experimental): Single ascending doses of ONO-7684 or placebo orally under fasted conditions
  Interventions: Drug: ONO-7684
- ONO-7684 Placebo Part A1 (Placebo Comparator): Single ascending doses of ONO-7684 or placebo orally under fasted conditions
  Interventions: Drug: ONO-7684 Placebo
- ONO-7684 Part A2 (Experimental): Single doses of ONO-7684 or placebo orally under fed conditions
  Interventions: Drug: ONO-7684
- ONO-7684 Placebo Part A2 (Placebo Comparator): Single doses of ONO-7684 or placebo orally under fed conditions
  Interventions: Drug: ONO-7684 Placebo
- ONO-7684 Part B1 (Experimental): Eligible subjects will receive multiple doses of ONO-7684 or placebo orally
  Interventions: Drug: ONO-7684
- ONO-7684 Placebo Part B1 (Placebo Comparator): Eligible subjects will receive multiple doses of ONO-7684 or placebo orally
  Interventions: Drug: ONO-7684 Placebo

INTERVENTIONS:
Drug: ONO-7684 — Single ascending doses for cohorts A1-A8 and multiple ascending doses cohorts B1-3
  Arms: ONO-7684 Part A1; ONO-7684 Part A2; ONO-7684 Part B1
Drug: ONO-7684 Placebo — Placebo comparator
  Arms: ONO-7684 Placebo Part A1; ONO-7684 Placebo Part A2; ONO-7684 Placebo Part B1

SUMMARY:
This is a first in human study to determine the safety, tolerability, pharmacokinetics and pharmacodynamics of ONO-7684 in healthy adult volunteers. This study will be conducted in 2 parts: Part A is a single-ascending dose and Part B is a multiple-ascending dose.

DETAILED DESCRIPTION:
This study aims to obtain safety, tolerability, pharmacokinetic and pharmacodynamic data when ONO-7684 is administered orally as single doses and as multiple doses to healthy subjects. The study will consist of 2 parts: A single ascending dose (SAD) phase (Part A); a multiple ascending dose (MAD) phase (Part B). One cohort of Part A will receive ONO-7684 under both fasted and fed conditions to investigate the effect of food.

ELIGIBILITY:
Inclusion Criteria:

1. 18-55 years
2. normotensive male volunteers, or female volunteers of non-childbearing potential (Part B only)
3. body mass index 18.0-30.0 kg/m2
4. deemed healthy on the basis of a clinical history, physical examination, ECG, vital signs, and laboratory tests of blood and urine
5. registered with a General Practitioner (GP) in the UK
6. agree to use an effective method of contraception
7. able to give fully informed written consent

Exclusion Criteria:

1. Positive tests for hepatitis B & C, HIV
2. severe adverse reaction to any drug
3. sensitivity to trial medication
4. drug or alcohol abuse
5. current smoker or use of nicotine containing products in the previous 6 months
6. vegetarians or vegans, or unwilling to eat a high-fat breakfast (Part A food effect cohorts only)
7. use of strong CYP3A4/5 or P-glycoprotein inhibitors or inducers, anticoagulants, antiplatelet agents, non-steroidal anti-inflammatory drugs and/or acetylsalicylic acid within the previous 30 days
8. prescription or over-the-counter medication, vitamins, herbal treatments or dietary supplements within the previous 7 days (with the exception of paracetamol [acetaminophen])
9. participation in other clinical trials of unlicensed medicines, or loss of more than 400 mL blood, within the previous 3 months or plan to donate blood or blood products in the 3 months after the trial
10. vital signs outside the acceptable range
11. clinically relevant abnormal findings at the screening assessment (including creatinine clearance, haemoglobin levels and QTcF)
12. acute or chronic illness
13. clinically relevant abnormal medical history or concurrent medical condition
14. objection by GP
15. possibility that volunteer will not cooperate
16. pre-menopausal females who are pregnant or lactating, or who are of childbearing potential

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 72 (Actual)
Dates: Start 2019-01-17 (Actual); Primary Completion 2019-08-23 (Actual); Study Completion 2019-08-23 (Actual)

PRIMARY OUTCOMES:
Number of participants with clinically significant changes in vital signs (Part A & B) | Part A: Day 1-4 & Follow-up and Part B: Day 1-15, 17 & Follow up
  Pulse rate (bpm), systolic and diastolic blood pressure (mmHg), Respiratory rate (bpm)
Number of participants with clinically significant changes observed on 12-lead electrocardiogram (ECG) (Part A & B) | Part A: Day 1-4 & Follow up & Part B: Day 1,3,5,7,9,11,14,17 & Follow up
  Ventricular rate (beats/min), PR interval (msec), QRS interval (msec), QT (msec), QTcF interval (msec)
Number of participants with clinically significant changes in cardiac telemetry (Part A only) | Part A: From 0.5-1 hours pre-dose until 12 hours after dosing at Day 1
  Number of participants with cardiac telemetry abnormalities will be reported.
Number of participants with clinically significant changes in physical examination (Part A & B) | Part A: Day -1, 1-4 & Follow-up and Part B: Day-1, 1-17 & Follow up
  Number of participants with physical examination abnormalities will be reported.
Number of participants with clinically significant changes in laboratory safety tests (haematology, biochemistry and urinalysis) (Part A & B) | Part A: Day-1, 1-4 & Follow up and Part B: Day-1, 1-17 & Follow up
  Number of participants with abnormalities in laboratory safety tests will be reported.
Number of participants with adverse events (AE) (Part A & B) | Part A: Day-1, 1-4 & Follow up and Part B: Day-1, 1-17 & Follow up
  AE is any untoward medical occurrence in a subject or clinical investigation subject, temporally associated with the use of a medicinal product, whether or not considered related to the medicinal product.

SECONDARY OUTCOMES:
Pharmacokinetics (Cmax) | Part A: Day 1 through Day 4. Part B: Day 1 and Day 14
  Assessment of the maximum observed plasma concentration of ONO-7684 and 3-hydroxybenzoic acid in Parts A and B
Pharmacokinetics (tmax) | Part A: Day 1 through Day 4. Part B: Day 1 and Day 14
  Assessment of the maximum observed plasma concentration of ONO-7684 and 3-hydroxybenzoic acid in Parts A and B
Pharmacokinetics (AUClast) | Part A: Day 1 through Day 4. Part B: Day 14
  Assessment of the area under the curve of ONO-7684 and 3-hydroxybenzoic acid in Parts A and B
Pharmacokinetics (AUCinf) | Part A: Day 1 through Day 4. Part B: Day 14
  Assessment of the area under the curve of ONO-7684 and 3-hydroxybenzoic acid in Parts A and B
Pharmacokinetics (AUCt) | Part A: Day 1 through Day 4. Part B: Day 1
  Assessment of the area under the curve of concentration of ONO-7684 and 3-hydroxybenzoic acid - time from zero up to a definitive time, t in Parts A and B
Pharmacokinetics (%AUCextrap) | Part A: Day 1 through Day 4. Part B: Day 14
  Assessment of the percentage of AUC∞ extrapolated from tlast to infinity of ONO-7684 and 3-hydroxybenzoic acid in Parts A and B
Pharmacokinetics (t1/2) | Part A: Day 1 through Day 4. Part B: Day 14
  Assessment of the elimination half-time of ONO-7684 and 3-hydroxybenzoic acid in Parts A and B
Pharmacokinetics (CL/F) | Day 1 through Day 4
  Assessment of the apparent clearance rate of ONO-7684 and 3-hydroxybenzoic acid in Part A only
Pharmacokinetics (Terminal Rate Constant) | Day 1 through Day 4
  Assessment of the terminal rate constant (slowest rate constant of the disposition) of ONO-7684 and 3-hydroxybenzoic acid in plasma in Part A only
Pharmacokinetics (Aet) | Day 1 through Day 4
  Assessment of the amount of ONO-7684 excreted in urine over the period of sample collection in Part A only
Pharmacokinetic (fe/F) | Day 1 through Day 4
  Assessment of the fraction of orally administered ONO-7684 excreted into urine in Part A only
Pharmacokinetic (CLr) | Day 1 through Day 4
  Assessment of the renal clearance of ONO-7684 from plasma in Part A only
Pharmacokinetic (Ctrough) | Day 1 through Day 14
  Assessment of the trough plasma concentration of ONO-7684 and 3-hydroxybenzoic acid in Part B only
Pharmacokinetic (AUCtau) | Day 14
  Assessment of the area under the plasma concentration of ONO-7684 and 3-hydroxybenzoic acid -time during a dosing interval in Part B only
Pharmacokinetic (CLSS/F) | Day 14
  Assessment of total clearance of ONO-7684 from plasma after oral administration in Part B only
Pharmacokinetic (VZ/F) | Day 14
  Assessment of apparent volume of distribution of ONO-7684 after non-intravenous administration calculated at steady state in Part B only
Pharmacodynamic (change from baseline in aPTT activity) in serum | Part A: Day 1 through Day 4. Part B: Day 1 through Day 17
  Assessment of the effect of ONO-7684 in activated partial thromboplastin time in Parts A and B
Pharmacodynamic (change from baseline in PT activity) in serum | Part A: Day 1 through Day 4. Part B: Day 1 through Day 17
  Assessment of the effect of ONO-7684 in prothrombin time in Parts A and B
Pharmacodynamic (change from baseline in PT-INR activity) in serum | Part A: Day 1 through Day 4. Part B: Day 1 through Day 17
  Assessment of the effect of ONO-7684 in prothrombin time-international normalised ratio in Parts A and B
Pharmacodynamic (change from baseline in FXIa activity) in serum | Part A: Day 1 through Day 4. Part B: Day 1 through Day 17
  Assessment of the effect of ONO-7684 in blood coagulation activated factor XI in Parts A and B
Pharmacodynamic (correlation of aPTT and FXIa activity) in serum | Part A: Day 1 through Day 4. Part B: Day 1 through Day 17
  Assessment of the effect of ONO-7684 in the correlation of activated partial thromboplastin time to blood coagulation activated factor XI in Parts A and B

CONTACTS AND LOCATIONS:
Locations (1):
- Hammersmith Medicines Research (HMR), London, United Kingdom